CLINICAL TRIAL: NCT05625516
Title: Bilateral External Torque CT, a Novel Diagnostic Tool for Detection of Syndesmotic Insufficiency
Status: Completed | Type: Observational
Sponsor: Balgrist University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-D0111
Record Dates: First submitted 2022-11-15; First posted 2022-11-23 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Syndesmotic Injuries
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with acute syndesmotic injuries: The patients undergo a bilateral external torque CT.
  Interventions: Device: Bilateral external torque device
- Patients with asymptomatic chronic syndesmotic injuries: The patients undergo a bilateral external torque CT.
  Interventions: Device: Bilateral external torque device
- Patients with symptomatic chronic syndesmotic injuries: The patients undergo a bilateral external torque CT.
  Interventions: Device: Bilateral external torque device

INTERVENTIONS:
Device: Bilateral external torque device — The "External Torque Device" was developed, which allows bilateral stressing of the syndesmosis by external rotation. Both lower legs are stabilized by a special knee brace (the fibula remains free to float) or by the hip joints, which are end rotated on both sides, while an external rotation force of maximum 7.5Nm (or up to the respective pain threshold) can be set on both sides using torque newton meters. If no load is possible - which the examination of the syndesmosis generally does not allow - an intra-articular local anesthesia with 5ml ropivacaine 2mg/ml can be performed under sterile conditions after the patient's consent.

SUMMARY:
Study population: the investigator set them sample size to 30 patients.

Primary endpoint (concerning both study questions): is the applied torque measurement in Newton meters (maximum up to 7.5 Nm) up to the pain tolerance limit. For the chronic injuries, a minimum of 5 Nm should be achieved. If this is not possible due to pain, an intra-articular infiltration into the upper ankle joint with 5ml Ropivacaine 2% is performed under sterile conditions.

In addition, fibula translation while exercising the maximum tolerated External Torque CT (maximum up to 7.5 Nm).

Secondary endpoint (1st study question): the comparison to stress fluoroscopy without anesthesia and under anesthesia.

Secondary endpoint (2nd study question): the comparison of patients with and without symptoms. Secondary endpoint in patients who received intra-articular infiltration is the increase in tolerated Newton meters.

DETAILED DESCRIPTION:
Isolated injuries to the distal tibiofibular syndesmosis affect approximately 1-17% of all ankle sprains and up to 30% in "high impact" sports. If the injury is missed, chronic syndesmosis instability can lead to prolonged convalescence, pain, and osteoarthritis of the upper ankle. Therefore, early diagnosis is essential for safe and effective treatment.

The diagnosis of syndesmosis insufficiency presents a certain dilemma in foot surgery. Already the differentiation between a simple fibular ligament lesion (low ankle sprain) and a syndesmosis injury (high ankle sprain) is often clinically difficult and only suggests a syndesmosis injury but does not confirm it.

The investigators have developed an external torque device that allows bilateral stressing of the syndesmosis by external rotation. In this case, both lower legs are stabilized by a special knee brace (fibula remains free floating) or by the hip joints, which are end rotated on both sides, while an external rotation force of maximum 7.5Nm (respectively up to the respective pain limit) can be set on both sides by means of torque newton meters. A CT can then be performed under external rotation stress.

In two previous studies (cadaver study and study on healthy subjects) the investigators have seen on the one hand that bilateral external torque CT is able to reliably detect syndesmosis instabilities and on the other hand that in healthy subjects the two ankle joints are comparable.

Based on these results the investigators want to address the following further questions:

1. can "Bilateral External Torque CT" be reliably applied in patients with acute syndesmosis rupture?
2. how stable does a syndesmosis have to be after an injury?

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Patient age of ≥18 yr and ≤75 yr.
* Proven acute (<4 weeks) syndesmosis injury (anterior and posterior) on MRI.
* Proven chronic (>2 months) syndesmosis injury (anterior and posterior) on MRI with/without surgical stabilization performed.
* Healthy opposite side

Exclusion Criteria:

* A dependency between patient sponsor and/or project management
* Pregnancy (contraindication for CT): in women of childbearing age, a pregnancy test is performed in any case
* St.n. previous operation(s) of the affected lower extremity (specifically of the ankle joint).
* Severe deformities (osteoarthritis with limited function upper and lower ankle joint, metatarsophalangeal joint).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 10 patients with acute syndesmotic injuries 10 patients with symptomatic chronic syndesmotic injuries 10 patients with aysmptomatic chronic syndesmotic injuries
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2023-08-31 (Actual); Primary Completion 2025-05-26 (Actual); Study Completion 2025-05-26 (Actual)

PRIMARY OUTCOMES:
External torque CT | 24 months
  = the applied torque measurement in Newton meters (maximum up to 7.5 Nm) up to the pain tolerance limit. In the chronic injuries, at least 5 Nm should be achieved. If this is not possible due to pain, patients with chronic injuries are infiltrated intra-articularly into the upper ankle joint with 5ml ropivacaine 2% under sterile conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Wirth, PD, Principal Investigator — Universitätsklinik Balgrist
Locations (1):
- Balgrist University Hospital, Zurich, Switzerland